CLINICAL TRIAL: NCT05752045
Title: Validation of OphtAI Software Diagnostic Performance for Automated Screening of Diabetic Retinopathy, Diabetic Macular Edema, Glaucoma, ARM and ARMD: a Multicentre Study
Brief Title: OphtAI Diagnostic Performance Validation for Automated Screening of Eye Diseases
Acronym: OPHTAI-EVAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evolucare Technologies (Industry)
Collaborators: Slb Pharma (Other); Assistance Publique - Hôpitaux de Paris (Other); BPIfrance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2022-A01813-40
Record Dates: First submitted 2023-01-25; First posted 2023-03-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema; Age-Related Macular Degeneration; Age-related Maculopathy; Glaucoma
Keywords: OphtAI; Artificial intelligence; Computer-aided diagnosis; Automated screening; Medical Device; Diabetic patient; Diabetic Retinopathy; Diabetic Macular Edema; Age-Related Macular Degeneration; Age-related Maculopathy; Glaucoma; Evolucare OphtAI
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration; Glaucoma

STUDY DESIGN:
Intervention Model Description: Imaging and clinical data will be collected from patients to be reviewed by an expert reader group providing ground truth, and the medical device will be tested against this ground truth
Masking Description: Ground truth and Results being obtained in the end of recruitment and imaging collection, there are no effects on participant or care provider. Also, experts won't be aware of AI results and vice versa.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetic patient group assessed for multiple eye diseases (Other): Each patient eye disease status will be assessed by expert readers so to provide ground truth against which algorithms performances will be assessed
  Interventions: Device: Eye Fundus Double Capture for Eye Diseases Screening with OphtAI Medical Device

INTERVENTIONS:
Device: Eye Fundus Double Capture for Eye Diseases Screening with OphtAI Medical Device — Double ophthalmological imaging capture of eye fundus with different fundus camera to screen patient for various eye diseases.

SUMMARY:
Evolucare OphtAI is a medical device offering automated, artificial intelligence powered, screening capabilities for Diabetic Retinopathy, Diabetic Macular Edema, Glaucoma, ARM and AMD, whose performances will by tested through the OphtAI-EVAL.

DETAILED DESCRIPTION:
OphtAI-Eval: is a prospective, multicentre, post-marketing clinical follow-up study (SCAC) of diagnostic validation (comparative vs gold standard).

It aims to: validate the diagnostic performance of the OphtAI software for the automated screening of diabetic retinopathy, diabetic macular edema, glaucoma, ARM and AMD.

Evolucare OphtAI is a medical imaging console for ophthalmology, interfaced with Evolucare Imaging.

It allows the detection, by statistical learning algorithms, of the following ocular pathologies using photographs of the retina:

* Diabetic retinopathy (DR) (including gradation),
* Diabetic macular edema (DME)
* Age-related macular degeneration (AMD)
* Age-related maculopathy (ARM, early form of AMD),
* Glaucoma.

Evolucare OphtAI, is available on the French market since March 2019.

ELIGIBILITY:
Doesn't not accept healthy volunteers as diabetic patients are needed, still they may be free of any eye diseases.

Inclusion Criteria:

The characteristics required for a subject to take part in the research are

* Male or female over 18,
* Type 1 or 2 diabetic,
* Presenting for screening for diabetic retinopathy,
* Beneficiary of a social security scheme,
* For whom written consent has been obtained for participation in the protocol.

Exclusion Criteria:

The following characteristics do not allow the subject to take part in the research:

* Patient with known DR, more severe than "minimal", including having been treated,
* Any other condition that, in the opinion of the health professionals, may interfere with their ability to complete the study or may present a significant risk,
* Presence of social, medical and/or psychological factors that may compromise the patient's adherence to the protocol,
* Simultaneously participating in another clinical research protocol or having recently participated in another research study for which the exclusion period would not be completed.

Patients who participate in this research will not be able to participate in another research at the same time. However, there is no exclusion period at the end of this research for participation in any other study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1389 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Referable Diabetic Retinopathy screening sensitivity/specificity | 1 year
  Referable Diabetic Retinopathy screening sensitivity/specificity evaluation (OphtAI software vs Expert reader) for RDR-EOphtha and RDR-OphDiaT_full algorithms

SECONDARY OUTCOMES:
Diabetic retinopathy grading sensitivity/specificity | 1 year
  Diabetic retinopathy grading performance (OphtAI software vs Expert reader) for each grading sub algorithms (sensitivity/specificity) and globally (accuracy/agreement ratio)
Diabetic retinopathy grading + RDR-EOphtha algorithms combination sensitivity/specificity for RDR detection | 1 year
  Referable Diabetic Retinopathy screening sensitivity/specificity evaluation (OphtAI software vs Expert reader) for RDR-EOphtha and RD grading algorithms combination
Diabetic retinopathy grading + RDR-OphDiaT_full algorithms combination sensitivity/specificity for RDR detection | 1 year
  Referable Diabetic Retinopathy screening sensitivity/specificity evaluation (OphtAI software vs Expert reader) for RDR-OphDiaT_full and RD grading algorithms combination
Diabetic retinopathy grading + RDR-EOphtha +DME algorithms combination sensitivity/specificity for RDR detection | 1 year
  Referable Diabetic Retinopathy screening sensitivity/specificity evaluation (OphtAI software vs Expert reader) for RDR-EOphtha, RD grading and DME algorithms combination
Diabetic retinopathy grading + RDR-OphDiaT_full +DME algorithms combination sensitivity/specificity for RDR detection | 1 year
  Referable Diabetic Retinopathy screening sensitivity/specificity evaluation (OphtAI software vs Expert reader) for RDR-OphDiaT_full , RD grading and DME algorithms combination
Diabetic Macular Edema algorithm sensitivity/specificityfor DME detection | 1 year
  Diabetic Macular Edema screening sensitivity/specificity evaluation (OphtAI software vs Expert reader) for DME algorithm
Age-Related Macular Degeneration algorithm sensitivity/specificity for AMD detection | 1 year
  AMD screening sensitivity/specificity evaluation (OphtAI software vs Expert reader) for AMD algorithm, for all forms and for either atrophic or neovascular AMD
Age-Related Maculopathy algorithm ("drusen") sensitivity/specificity for ARM detection | 1 year
  ARM screening sensitivity/specificity evaluation (OphtAI software vs Expert reader) for ARM algorithm, for all forms and for either macular or peripheric drusen, or for either hard/soft drusen
Glaucoma algorithms sensitivity/specificity for Glaucoma suspicion | 1 year
  Glaucoma screening sensitivity/specificity evaluation (OphtAI software vs Expert reader) for Glaucoma algorithms
Quality algorithm accuracy for quality assessment | 1 year
  Bad quality images sensitivity/specificity evaluation (OphtAI software vs Expert reader) for quality assessment algorithms
Laterality determination algorithm accuracy for laterality assessment | 1 year
  Laterality accuracy of OphtAI software vs Expert reader for laterality determination algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Aude Couturier, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (12):
- France (12):
  - Centre Aix Vision, Aix-en-Provence
  - CHU Brest, Brest
  - Centre Ophtalmologique Brétigny Essonne, Brétigny-sur-Orge
  - CH SUD Francilien Corbeil Essonne, Corbeil-Essonnes
  - Centre d'examens de santé de la CPAM 93, Corbeil-Essonnes
  - Retinodiab Bourgogne, Dijon
  - Clinique Honoré Cave, Montauban
  - CHU Nantes, Nantes
  - Retinodiab Franche-Comté, Roppe
  - Diabète Occitanie, Toulouse
  - CHU Toulouse, Toulouse
  - OPHDIAT, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No